CLINICAL TRIAL: NCT01418170
Title: Dose Response Effects of Cervical SMT on Pressure Sensitivity of Myofascial Trigger Points
Brief Title: Dose Response Effects of Cervical Spinal Manipulative Therapy (SMT) on Pressure Sensitivity of Myofascial Trigger Points
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Memorial Chiropractic College (Other)
Collaborators: University of Guelph (Other)
Responsible Party: Dr. Michelle Laframboise, Canadian Memorial Chiropractic College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 112027
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2011-08

CONDITIONS: Trigger Points, Myofascial; Myofascial Trigger Points; Myofascial Pain Syndrome
Keywords: myofascial pain syndrome; myofascial trigger points; spinal manipulative therapy; algometer; pressure pain thresholds
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Two rcSMT group (Experimental): A rcSMT will be performed to the C5-C6 segment. A thrust maneuver will then be given to the C5-C6 segment. A rotational inferior drop thrust maneuver will be performed. Immediately after the first rcSMT the subject will turn over on the chiropractic table to lie in the prone position for a post-rcSMT PPT measurement with the same algometer performed by the research assistant. These will be taken at 5-minute intervals. A second rcSMT will be performed at 30 minutes after the first rcSMT. The invention protocol will be repeated. The subject will turn over to the prone position for repeat PPT measurements at 5-minute intervals post-rcSMT for 30 mins. Once the subject has left the treatment area the clinician will mark on the treatment card whether the rcSMT was performed with or without cavitation for quality control purposes.
  Interventions: Other: cervical spinal manipulative therapy
- One scSMT + One rcSMT Group (Sham Comparator): A scSMT will be performed with the contact hand of the clinician resting lightly on the paraspinal area of the neck of the subject. The subject's head will be rotated to 45 degrees and supported by the clinician's forearm, lying on headpiece. A inferior drop thrust will be applied to the drop piece. After the first scSMT maneuver the subject will turn over on the chiropractic table to lie in the prone position for a post-scSMT PPT measurement. PPT measurements will be taken at 5-minute intervals for 30 minutes. A rcSMT will be performed 30 minutes after the first scSMT. The subject will turn over to the prone position for repeat PPT measurements in 5-minute intervals for 30 minutes post-rcSMT. Once the subject has left the treatment area the clinician will mark on the treatment card weather the scSMT was performed adequately without cavitation and whether a cavitation occurred with the rcSMT.
  Interventions: Other: cervical spinal manipulative therapy

INTERVENTIONS:
Other: cervical spinal manipulative therapy — A real cervical spine manipulation will be used for the intervention vs a sham cervical spine manipulation. For the rcSMT the subject's head will be supported by the clinician's forearm. The contact hand of the clinician will contact the C5-C6 spinal segment. A thrust maneuver will be given by the contact hand of the clinician with the supportive hand resting on the subject's zygoma. A rotational inferior drop thrust maneuver will be completed. For the scSMT the subject's head will be rotated to 45 degrees and will be supported by the clinician's forearm, which will lie on top if the headpiece. A thrust maneuver will then be given by the contact hand of the treating clinician to the drop piece with the hand beside the paraspinal musculature simulating a real thrust, the supportive hand will be resting on the subject's zygoma. A inferior drop thrust will be applied to the drop piece (no thrust is made by the contact hand on the cervical spine).

SUMMARY:
Specific Aim 1:

To determine if the effect of cervical spinal manipulation on the pressure pain thresholds in a myofascial trigger point in the infraspinatus muscle can be enhanced and/or extended after a second cervical spine manipulation is given during a single subject visit.

H1: There will be a statistically significant increase in pressure pain thresholds in the myofascial trigger point in the infraspinatus muscle after the second cervical spine manipulation, as compared to the first.

Specific Aim 2:

To determine if the effect of two cervical spinal manipulations on pressure pain thresholds in a myofascial trigger point in the infraspinatus muscle will be present at 48 hours follow-up. Data will be collected for descriptive purposes and hypothesis generation.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is one of the most common manifestations of myofascial pain syndromes. The total annual cost of FMS is $2298 per patient in Canada. A Canadian study suggests that FMS-related productivity loss costs per year are $10,068 per patient. The average cost of health resources in Canada is 30% higher in FMS patients compared to non-FMS patients and the prevalence of FMS in Canada is 1.1%, leading to a total of over 340 thousand Canadians suffering from FMS. As a result, the annual economic burden of FMS to the Canadian healthcare system is more than $425 million.

Typically, FMS patients have widespread musculoskeletal pain with associated non-specific tender points. There is an increase in prevalence in active myofascial trigger points (MTrPs) contributing to the widespread musculoskeletal pain associated with FMS patients. MTrPs are identified as hyperirritable muscular nodules located within taut bands of skeletal muscle and can be classified as latent or active. Studies have shown that active and latent MTrPs can play a determinant role in the not yet fully understood pathogenesis of FMS.

There are many common pathophysiological theories that exist for MTrP formation including metabolic, biochemical, motor endplate dysfunction, and the neurogenic phenomenon. MTrPs may be initiated by a sensitization within the common neurologic segment of the specific tissue containing the MTrP. The physiological changes that occur at the MTrP are secondary to an increased responsiveness of the neurons within the central nervous system leading to increased nociception and increased perception of pain.

Currently there are a variety of therapeutic techniques established to treat MTrPs including spinal manipulative therapy (SMT). SMT may attenuate the nociceptive component of spinal pain and MTrPs. SMT increases pressure pain thresholds (PPTs) leading to mechanical hypoalgesia of MTrPs in paraspinal muscles. Preliminary data collected by Srbely et al. has shown that there is a significant increase in PPTs in infraspinatus MTrPs after cSMT to the C5-C6 spinal segments compared to a sham procedure. The measure of PPT is a method of quantifying a patient's perception of pain in a MTrP. PPTs can be defined as the least amount of pressure stimulus at which a subject perceives pain upon the application of pressure in the form of force.

The appropriate dosage (frequency of application) of SMT needed to achieve optimal pain relief for patients with MTrPs has not been established. Haas et al. performed a pilot randomized controlled trial to examine the dose response relationship between SMT and cervicogenic headaches. The results showed there is a dose-response relationship, increasing the dose of SMT leads to a decreased frequency and intensity of headaches. Additionally, Haas and colleagues conducted a pilot study to make a preliminary identification of the number of chiropractic manipulations required to decrease chronic low back pain and disability. The results showed a positive dose-response relationship between SMT and low back pain. Dose-response for MTrPs has yet to be established in the current literature. This preliminary work will determine the proper dose-response for cSMT in the treatment of MTrPs in one single visit.

Specific Aim 1:

To determine if the effect of cervical SMT on the PPT in a MTrP in the infraspinatus muscle can be enhanced and/or extended after a 2nd cSMT is given during a single subject visit.

H1: There will be a statistically significant increase in PPTs in the MTrP in the infraspinatus muscle after the second cervical SMT, as compared to the first.

Specific Aim 2:

To determine if the effect of two cervical SMTs on PPTs in a MTrP in the infraspinatus muscle will be present at 48 hours follow-up. Data will be collected for descriptive purposes and hypothesis generation.

Studies show that manual therapy including SMT, is a cost effective method for treating chronic pain and FMS. Currently, treatment protocols are arbitrarily selected based on opinion or clinical experience. Providing proper guidelines for MTrP and SMT can increase the effectiveness of treatment plans and decrease the financial cost of FMS on patients and the healthcare system. For this preliminary work, looking at MTrP mechanism is best done in isolation of FMS and therefore subjects without FMS will be used.

Recruitment Process Subjects will be recruited via convenience sampling from the Canadian Memorial Chiropractic College campus and main campus clinic through announcements, advertising, educating the student body and clinicians on the specific aims of this particular study, by emailing the student body asking for volunteers, and by direct recruitment through personal contact

Subject Screening The research assistant will assess all volunteers for eligibility. The demographics of all of the volunteers will be collected including gender, age, height, weight, hand dominance, and ethnicity. Demographics will be collected so that this information can be compared to subjects that do have MTrPs in the infraspinatus muscle. All volunteers meeting the eligibility criteria will be included. Reasons for exclusion will be collected. Eligible healthy subjects will move on to a physical examination of the cervical spine. The physical assessment will include a cervical range of motion screen, palpation of the cervical spine, palpation of the infraspinatus muscle bilaterally, and an upper limb neurological examination. Documentation if there was pain on palpation of the infraspinatus MTrP occurred, if there was referral to the lateral aspect of the shoulder with or without palpation of the infraspinatus MTrP, and if there was a local twitch response in the infraspinatus MTrP for baseline information. Documentation if the MTrP is active or latent will be performed at baseline and if there is failure of randomization a statistical analysis will be performed. If, during the assessment the subject reports pain with cervical range of motion, or cervical palpation, the presence of arm pain, decreased motor examination, abnormal sensation, or the presence of hyper-reflexia or hypo-reflexia, the examination will be terminated and the subject will be excluded from the study. Subjects with a MTrP in the infraspinatus muscle will have a baseline PPT measurement performed with an algometer to ensure the MTrP meets the inclusion of no more than 35N. Subjects that have no cervical spine pain, no arm pain, and no neurological symptoms and a MTrP in the infraspinatus muscle no more than 35N will be included in the study.

Those included in the study will be randomly allocated to two separate groups. A predetermined computer generated random allocation sequence will be used to separate individuals into two groups, those who receive two rcSMT and those who receive one rcSMT and one scSMT. The statistician will hold the randomization scheme. To ensure proper concealment the statistician will not be involved in the experiment and the clinician and research assistant will not be involved in the randomization scheme. The individual group allocations will be printed by the research assistant and placed into blank white opaque numbered envelopes. The white opaque envelopes will be numbered 001→ 013 for males and 014→026 for females. The research assistant will record the number from the envelope on the subject information sheet. The research assistant will give the participant an envelope to give to the clinician. The research assistant will be blinded but the clinician will be educated what the codes mean. The clinician will open the opaque numbered envelope and discretely look at the randomization scheme printed on the white card inside, ensuring that the subject does not see the randomization scheme. The card with the randomization scheme on it will then be placed back in the opaque numbered envelope. For quality control purposes cavitation of the rcSMT and scSMT will be monitored by the clinician, any cavitation in the scSMT will be documented and accounted for.

Compensation The participants will receive compensation totaling $35.00 in the form of two Tim Horton's gift cards (one for 10 dollars one for 25 dollars) in recognition of the subject's time, parking, and gasoline. Subjects will receive a 5-dollar gift card if they volunteer and are found not to have a MTrP in the infraspinatus muscle. A 10-dollar gift card will be provided to those that complete the first day of the experiment and 25-dollar gift card will be provided to those that follow-up after 48 hours.

Methods related to both Specific Aims Eligible subjects will be asked to first read an information letter and then sign an informed consent form for cSMT after all questions are answered prior to the physical examination. The research assistant will then give the subjects a gown to change into, all clothes covering the upper thorax, abdomen, and upper extremities must be removed including but not limited to earrings, necklaces, bras, undershirts, t-shirts, and sweaters. The subjects will be instructed by the research assistant to place the gown on with the ties facing the back to facilitate palpation of the infraspinatus muscle. Subjects will then be instructed to enter the lab and lie prone on the chiropractic table. A black non-toxic marker will be used to indicate the exact location of the MTrP in the infraspinatus muscle. The baseline PPT of the infraspinatus muscle will be taken with a handheld algometer by the research assistant. For reliability PPT measures will be taken 3 consecutive times at each time point. Following the baseline procedures, subjects will move into the supine position on the chiropractic table with the head on a drop piece. The clinician will be at the end of the chiropractic table where the subject's head will rest on the drop headpiece. The clinician will perform either an intervention of two consecutive rcSMT or one scSMT followed by one rcSMT on the ipsilateral side of the infraspinatus MTrP. Manipulation of the cervical spine will be applied to the C5-C6 segments with a force indicated for gapping the joint. After the intervention each subject will be asked to fill out a questionnaire to address subject treatment expected bias. The subjects will fill out the questionnaire and place it in a sealed numbered envelope and give it to the research assistant. Prior to leaving all subjects will be reminded by the research assistant to retrain from any musculoskeletal treatments or use of any medications not previously prescribed.

Specific Aim #1

Two rcSMT Group:

A rcSMT will be performed contacting the C5-C6 segment. The subject's head will be supported by the clinician's forearm. The contact hand of the clinician will contact the C5-C6 spinal segment. A thrust maneuver will then be given by the contact hand of the clinician to the C5-C6 segment with the supportive hand resting on the zygoma of the subject. A rotational inferior drop thrust maneuver will be completed19. Immediately after the first rcSMT the subject will turn over on the chiropractic table to lie in the prone position for a post-rcSMT PPT measurement with the same algometer performed by the research assistant. This post-rcSMT PPT measurement will be taken at 5-minute intervals after the first rcSMT. Once the PPT measurement is taken the subject will be asked to rest quietly in the supine position with the head resting on the drop headpiece. A second rcSMT will be performed at 30 minutes after the first rcSMT. The same invention protocol will be repeated. Successive rcSMT will be 30 minutes part based on the results from Ross et al. showing that a second cavitation of the same joint cannot occur before 20 minutes. Thus, 30 minutes will be used so that another cavitation of the C5-C6 segment is possible with a 10-minute buffer to account for any possible technical difficulties. The subject will turn over to the prone position for repeat PPT measurements at 5-minute intervals post-rcSMT for 30 mins. Once the PPT measurements are taken the subject will be free to leave and will be compensated. Once the subject has left the treatment area the clinician will mark on the treatment card whether the rcSMT was performed with or without cavitation for quality control purposes and place the treatment card back in its specified numbered envelope and drop it in a drop box that will be place in the treatment area.

One scSMT + One rcSMT Group A scSMT will be performed with the contact hand of the clinician resting lightly on the paraspinal area of the neck of the subject. The subject's head will be rotated to 45 degrees and will be supported by the clinician's forearm, which will lie on top if the headpiece. A thrust maneuver will then be given by the contact hand of the treating clinician to the drop piece with the hand beside the paraspinal musculature simulating a real thrust, the supportive hand will be resting on the zygoma of the subject. A inferior drop thrust will be applied to the drop piece (no thrust is made by the contact hand on the cervical spine) (Figure 3 and 4)19. Immediately after the first scSMT maneuver the subject will turn over on the chiropractic table to lie in the prone position for a post-scSMT PPT measurement with the same algometer performed by the research assistant. This post-scSMT PPT measurement will be taken at 5-minute intervals for 30 minutes after the first scSMT. A rcSMT will be performed 30 minutes after the first scSMT. The subject will turn over to the prone position for repeat PPT measurements in 5-minute intervals for 30 minutes post-rcSMT. Once the PPT measurement is taken the subject will be free to leave the treatment area. Once the subject has left the treatment area the clinician will mark on the treatment card weather the scSMT was performed adequately without cavitation and whether a cavitation occurred with the rcSMT or not and place the treatment card back in its specified numbered envelope and drop it in a drop box that will be place in the treatment area.

Specific Aim #2 All subjects regardless of the group will be required to attend a 48-hour follow-up after the intervention. The purpose of the follow-up will be to determine the how long the effect of the cSMT will last on PPT measurements taken on the infraspinatus MTrP. Subjects will be called for a follow-up reminder by the research assistant 1 day prior to follow-up to increase compliance. Subjects will present to the Canadian Memorial Chiropractic College and will be greeted by the same research assistant (See Specific Aim #1 methods). The permanent black mark will be identified for proper infraspinatus MTrP PPT measurement. A permanent black will be used to ensure same MTrP will be measured to set the same scene as 48 hours prior to follow-up. The research assistant will then take one PPT measurement with a handheld algometer on the same MTrP. The subjects will be asked to change back into clothing and provided with compensation.

Blinding and Minimization of Bias This study will be a single-blinded RCT in that the subjects, statistician providing the randomization scheme, and the research assistant performing the physical examination will all be blinded. The experienced clinician providing the rcSMT or scSMT procedure will not be blinded. The experienced clinician will have to know which group the subject is in to be able to perform the proper intervention (two rcSMT or one scSMT and one rcSMT). The bias in administering the SMT intervention in this study will be minimized by employing a validated sham procedure created by Vernon et al. in 2005. The subject treatment expected bias will be accounted for by recording patient perceptions of the treatment protocol.

Compliance and Co-intervention For the primary specific aim of this study compliance will not be a problem due to the limited time needed for the experiment. Compliance for the secondary aim where a 2-day follow-up is required for data collection may be more challenging. However, the follow-up will be very short consisting of one PPT measurement with a hand held algometer. Thus, the time requirement will be approximately 10 minutes in length. Further, subjects involved in the experiment will be students and faculty at the Canadian Memorial Chiropractic College the same institution that data collection will occur making the follow-up more convenient for subjects. Compliance will be increased by a phone call made by the research assistant to the subject one day prior to follow-up for a friendly reminder. Also, a gift card will be given out upon study completion to increase subject compliance. Co-intervention will be avoided by employing the specified eligibility criteria. Co-intervention will be avoided due to the short time span of the experimental maneuver. Study participates cannot have had any SMT in the pervious month. This washout period of treatment is needed to avoid co-intervention. Subjects will be instructed not to have any manual treatment between the experiment and the 48-hour follow-up to avoid co-intervention. If treatment of the cervical spine occurs data analysis will be modified to account for this. Documentation if treatment occurred between intervention and follow-up will be used to see if there is a significant outcome from non-compliance.

Analysis A 2F repeated measures ANOVA will be performed using STATA version 11 software (StataCorp LP, College Station, Texas, USA). The within groups analysis will look at time points and the between groups analysis will look at group differences. A Post Hoc analysis will be performed. All raw PPT measures will be normalized to baseline to account for subject variability. A statistician will be conducting the data analysis with the STATA software. Descriptive statistics will be used for the secondary aim of this study.

ELIGIBILITY:
Inclusion Criteria:

* female subjects between the ages of 21-40 from the Canadian Memorial Chiropractic College (CMCC) main campus and campus clinic
* MTrPs in the infraspinatus muscle

Exclusion Criteria:

* Received cSMT within the 72 hour*
* Insufficient English language to complete pre-study questionnaires
* No MTrP in the infraspinatus muscle
* PPT in the MTrPs in the infraspinatus of greater than 35N
* Any absolute or relative contraindications to manipulation such as; previous VBI, blood-clotting disorders, hypertension, or cardiovascular disorders
* Any current or prior history of neurological signs and symptoms including facial or extremity weakness, abnormal sensation to the face, body, upper, or lower extremities, uncontrolled bodily movements, gait disturbances, unexplained dizziness, unexplained nausea or vomiting, difficulty with speaking or swallowing
* Previous history of a whiplash associated disorder
* Previous cervical spine surgery
* Any current or recent cervical or thoracic injury including cervical disc herniation with or without radiculopathy, facet irritation, fracture to the cervical spine, fracture to the thoracic spine, or fracture to the scapula
* Concomitant injuries and/or co-morbidities affecting the cervical, thoracic, upper limb musculoskeletal system and systemic diseases affecting the musculoskeletal system such as diabetes, muscular dystrophies, or chronic pain disorders
* Current nerve entrapments in the upper extremities
* Myositis ossificans in the infraspinatus muscle
* Seronegative spondyloarthropathies
* Current use of medications such as NSAIDS, antidepressants, or opioids *A wash out period of no cSMT is needed because people accommodate to treatment. A 72-hour time period was chosen as it allows sufficient time for any effects of cSMT on MTrPs to disappear

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change scores of the pressure algometry | 5 minute intervals for 30 minutes post SMT
  The outcome being measured is PPTs of MTrP in the infraspinatus muscle with a digital hand-held algometer. PPT readings will be recorded in Newtons, the amount of force required to accelerate a 1-kg mass at 1m/s. MTrP with a baseline PPT of 35N or less will be included. PPT readings will be taken with a hand-held force gauge (NexGen Chatillon DFE Series, AMETEK TCI, Florida, USA) the force gauge tip will be 285mm2 (19 mm x 15 mm). PPT readings will be taken with a force gauge by applying a progressive increase in force perpendicular to the skin at the rate of 5N/s over the MTrP.

SECONDARY OUTCOMES:
Change scores of the pressure algometry | 5 minutes
  A follow-up pressure pain score will be taken by a pressure algometer 48 hours after the initial intervention.
The perception by subjects as to whether they received a real treatment | 5 minutes
  After the intervention the subjects will be asked whether they received a real cSMT or the sham cSMT.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A Laframboise, BKin (Hons), DC, Principal Investigator — Canadian Memorial Chiropractic College
Locations (1):
- Canadian Memorial Chiropractic College, Toronto, Ontario, Canada

REFERENCES:
- [Background] Scott NA, Guo B, Barton PM, Gerwin RD. Trigger point injections for chronic non-malignant musculoskeletal pain: a systematic review. Pain Med. 2009 Jan;10(1):54-69. doi: 10.1111/j.1526-4637.2008.00526.x. Epub 2008 Nov 5. PMID 18992040
- [Background] Meyer HP. Myofascial pain syndrome and its suggested role in the pathogenesis and treatment of fibromyalgia syndrome. Curr Pain Headache Rep. 2002 Aug;6(4):274-83. doi: 10.1007/s11916-002-0048-z. PMID 12095462
- [Background] Penrod JR, Bernatsky S, Adam V, Baron M, Dayan N, Dobkin PL. Health services costs and their determinants in women with fibromyalgia. J Rheumatol. 2004 Jul;31(7):1391-8. PMID 15229962
- [Background] Lachaine J, Beauchemin C, Landry PA. Clinical and economic characteristics of patients with fibromyalgia syndrome. Clin J Pain. 2010 May;26(4):284-90. doi: 10.1097/AJP.0b013e3181cf599f. PMID 20393262
- [Background] Ge HY, Nie H, Madeleine P, Danneskiold-Samsoe B, Graven-Nielsen T, Arendt-Nielsen L. Contribution of the local and referred pain from active myofascial trigger points in fibromyalgia syndrome. Pain. 2009 Dec 15;147(1-3):233-40. doi: 10.1016/j.pain.2009.09.019. Epub 2009 Oct 9. PMID 19819074
- [Background] Ge HY, Wang Y, Danneskiold-Samsoe B, Graven-Nielsen T, Arendt-Nielsen L. The predetermined sites of examination for tender points in fibromyalgia syndrome are frequently associated with myofascial trigger points. J Pain. 2010 Jul;11(7):644-51. doi: 10.1016/j.jpain.2009.10.006. Epub 2009 Nov 14. PMID 19914876
- [Background] Ge HY. Prevalence of myofascial trigger points in fibromyalgia: the overlap of two common problems. Curr Pain Headache Rep. 2010 Oct;14(5):339-45. doi: 10.1007/s11916-010-0127-5. PMID 20607459
- [Background] Alonso-Blanco C, Fernandez-de-las-Penas C, Morales-Cabezas M, Zarco-Moreno P, Ge HY, Florez-Garcia M. Multiple active myofascial trigger points reproduce the overall spontaneous pain pattern in women with fibromyalgia and are related to widespread mechanical hypersensitivity. Clin J Pain. 2011 Jun;27(5):405-13. doi: 10.1097/AJP.0b013e318210110a. PMID 21368661
- [Background] Simons DG. Review of enigmatic MTrPs as a common cause of enigmatic musculoskeletal pain and dysfunction. J Electromyogr Kinesiol. 2004 Feb;14(1):95-107. doi: 10.1016/j.jelekin.2003.09.018. PMID 14759755
- [Background] Srbely JZ. New trends in the treatment and management of myofascial pain syndrome. Curr Pain Headache Rep. 2010 Oct;14(5):346-52. doi: 10.1007/s11916-010-0128-4. PMID 20607458
- [Background] Majlesi J, Unalan H. Effect of treatment on trigger points. Curr Pain Headache Rep. 2010 Oct;14(5):353-60. doi: 10.1007/s11916-010-0132-8. PMID 20652653
- [Background] Fernandez-de-Las-Penas C, Ge HY, Arendt-Nielsen L, Cuadrado ML, Pareja JA. Referred pain from trapezius muscle trigger points shares similar characteristics with chronic tension type headache. Eur J Pain. 2007 May;11(4):475-82. doi: 10.1016/j.ejpain.2006.07.005. Epub 2006 Aug 21. PMID 16919982
- [Background] Fernandez-de-Las-Penas C, Alonso-Blanco C, Cleland JA, Rodriguez-Blanco C, Alburquerque-Sendin F. Changes in pressure pain thresholds over C5-C6 zygapophyseal joint after a cervicothoracic junction manipulation in healthy subjects. J Manipulative Physiol Ther. 2008 Jun;31(5):332-7. doi: 10.1016/j.jmpt.2008.04.006. PMID 18558274
- [Background] Vernon HT, Aker P, Burns S, Viljakaanen S, Short L. Pressure pain threshold evaluation of the effect of spinal manipulation in the treatment of chronic neck pain: a pilot study. J Manipulative Physiol Ther. 1990 Jan;13(1):13-6. PMID 2324655
- [Background] Vernon H. Qualitative review of studies of manipulation-induced hypoalgesia. J Manipulative Physiol Ther. 2000 Feb;23(2):134-8. doi: 10.1016/s0161-4754(00)90084-8. PMID 10714544
- [Background] Vernon H, MacAdam K, Marshall V, Pion M, Sadowska M. Validation of a sham manipulative procedure for the cervical spine for use in clinical trials. J Manipulative Physiol Ther. 2005 Nov-Dec;28(9):662-6. doi: 10.1016/j.jmpt.2005.07.020. PMID 16326235
- [Background] Haas M, Spegman A, Peterson D, Aickin M, Vavrek D. Dose response and efficacy of spinal manipulation for chronic cervicogenic headache: a pilot randomized controlled trial. Spine J. 2010 Feb;10(2):117-28. doi: 10.1016/j.spinee.2009.09.002. PMID 19837005
- [Background] Haas M, Groupp E, Kraemer DF. Dose-response for chiropractic care of chronic low back pain. Spine J. 2004 Sep-Oct;4(5):574-83. doi: 10.1016/j.spinee.2004.02.008. PMID 15363431
- [Background] Groeneweg R, Kropman H, Leopold H, van Assen L, Mulder J, van Tulder MW, Oostendorp RA. The effectiveness and cost-evaluation of manual therapy and physical therapy in patients with sub-acute and chronic non specific neck pain. Rationale and design of a Randomized Controlled Trial (RCT). BMC Musculoskelet Disord. 2010 Jan 24;11:14. doi: 10.1186/1471-2474-11-14. PMID 20096136
- [Background] Vernon H, Humphreys BK. Manual therapy for neck pain: an overview of randomized clinical trials and systematic reviews. Eura Medicophys. 2007 Mar;43(1):91-118. PMID 17369783
- [Background] Vernon H, Humphreys K, Hagino C. Chronic mechanical neck pain in adults treated by manual therapy: a systematic review of change scores in randomized clinical trials. J Manipulative Physiol Ther. 2007 Mar-Apr;30(3):215-27. doi: 10.1016/j.jmpt.2007.01.014. PMID 17416276
- [Background] Hurwitz EL, Carragee EJ, van der Velde G, Carroll LJ, Nordin M, Guzman J, Peloso PM, Holm LW, Cote P, Hogg-Johnson S, Cassidy JD, Haldeman S; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Treatment of neck pain: noninvasive interventions: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S123-52. doi: 10.1097/BRS.0b013e3181644b1d. PMID 18204386
- [Background] Srbely JZ, Dickey JP, Bent LR, Lee D, Lowerison M. Capsaicin-induced central sensitization evokes segmental increases in trigger point sensitivity in humans. J Pain. 2010 Jul;11(7):636-43. doi: 10.1016/j.jpain.2009.10.005. Epub 2009 Dec 16. PMID 20015704
- [Background] Srbely JZ, Dickey JP, Lee D, Lowerison M. Dry needle stimulation of myofascial trigger points evokes segmental anti-nociceptive effects. J Rehabil Med. 2010 May;42(5):463-8. doi: 10.2340/16501977-0535. PMID 20544158
- [Background] Vanderweeen L, Oostendorp RA, Vaes P, Duquet W. Pressure algometry in manual therapy. Man Ther. 1996 Dec;1(5):258-265. doi: 10.1054/math.1996.0276. PMID 11440515
- [Background] Fischer AA. Pressure algometry over normal muscles. Standard values, validity and reproducibility of pressure threshold. Pain. 1987 Jul;30(1):115-126. doi: 10.1016/0304-3959(87)90089-3. PMID 3614975
- [Background] Antonaci F, Sand T, Lucas GA. Pressure algometry in healthy subjects: inter-examiner variability. Scand J Rehabil Med. 1998 Mar;30(1):3-8. doi: 10.1080/003655098444255. PMID 9526748
- [Background] Ylinen J, Nykanen M, Kautiainen H, Hakkinen A. Evaluation of repeatability of pressure algometry on the neck muscles for clinical use. Man Ther. 2007 May;12(2):192-7. doi: 10.1016/j.math.2006.06.010. Epub 2006 Sep 7. PMID 16956783
- [Background] Kinser AM, Sands WA, Stone MH. Reliability and validity of a pressure algometer. J Strength Cond Res. 2009 Jan;23(1):312-4. doi: 10.1519/jsc.0b013e31818f051c. PMID 19130648
- [Background] Chesterton LS, Sim J, Wright CC, Foster NE. Interrater reliability of algometry in measuring pressure pain thresholds in healthy humans, using multiple raters. Clin J Pain. 2007 Nov-Dec;23(9):760-6. doi: 10.1097/AJP.0b013e318154b6ae. PMID 18075402
- [Background] Skootsky SA, Jaeger B, Oye RK. Prevalence of myofascial pain in general internal medicine practice. West J Med. 1989 Aug;151(2):157-60. PMID 2788962
- [Background] Assendelft WJ, Bouter LM, Knipschild PG. Complications of spinal manipulation: a comprehensive review of the literature. J Fam Pract. 1996 May;42(5):475-80. PMID 8642364
- [Background] Hurwitz EL, Morgenstern H, Vassilaki M, Chiang LM. Adverse reactions to chiropractic treatment and their effects on satisfaction and clinical outcomes among patients enrolled in the UCLA Neck Pain Study. J Manipulative Physiol Ther. 2004 Jan;27(1):16-25. doi: 10.1016/j.jmpt.2003.11.002. PMID 14739870
- [Background] Staud R. Future perspectives: pathogenesis of chronic muscle pain. Best Pract Res Clin Rheumatol. 2007 Jun;21(3):581-96. doi: 10.1016/j.berh.2007.02.013. PMID 17603001
- [Background] Pickar JG. Neurophysiological effects of spinal manipulation. Spine J. 2002 Sep-Oct;2(5):357-71. doi: 10.1016/s1529-9430(02)00400-x. PMID 14589467
- [Background] Pickar JG. An in vivo preparation for investigating neural responses to controlled loading of a lumbar vertebra in the anesthetized cat. J Neurosci Methods. 1999 Jul 15;89(2):87-96. doi: 10.1016/s0165-0270(99)00060-6. PMID 10491938
- [Background] Terrett AC, Vernon H. Manipulation and pain tolerance. A controlled study of the effect of spinal manipulation on paraspinal cutaneous pain tolerance levels. Am J Phys Med. 1984 Oct;63(5):217-25. PMID 6486245